CLINICAL TRIAL: NCT04432285
Title: Long-term Outcome in Cervical Dystonia Patients Treated With Chronic Pallidal Deep Brain Stimulation Compared to Repeated Botulinum Toxin Injections - a Cross-sectional Observational Study
Brief Title: Long-term Outcome of DBS Versus Botulinum Toxin Treatment in Cervical Dystonia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Inger Marie Skogseid, Consultant neurologist, Project leader, Oslo University Hospital
Other Study IDs: 96307
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Cervical Dystonia
Keywords: Deep Brain Stimulation; Botulinum Toxin treatment
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deep Brain Stimulation (GPi-DBS): Patients with cervical dystonia (CD) who were operated at Oslo University Hospital between June 2004 and December 2017 with a DBS-device targeting the GPi bilaterally, and who have been treated with chronic GPi-DBS for a minimum of 3 years.
  Interventions: Device: DBS-device, implanted in GPi bilaterally
- Botulinum toxin treatment: CD patients who for a minimum of 3 years have received treatment with botulinum neurotoxin (BoNT) injections at regular intervals (minimum 12 injection cycles) and still are receiving them (Age- and gender matched to the GPi-DBS group)
  Interventions: Drug: Botulinum toxin

INTERVENTIONS:
Device: DBS-device, implanted in GPi bilaterally — Chronic/continuous bilateral GPi-DBS
  Groups: Deep Brain Stimulation (GPi-DBS)
Drug: Botulinum toxin — Repeated intramuscular injections at regular intervals of around 3 months
  Groups: Botulinum toxin treatment

SUMMARY:
Cervical dystonia (CD) is the most common isolated dystonia in adults. Cervical dystonia symptoms can in most patients be managed well by botulinum toxin (BTX) injections, and supporting treatment measures. However, one-fifth to one-third of patients do not obtain sufficient relief from long-term BTX therapy, resulting in reduced quality of life. Deep brain stimulation (DBS) is a treatment method in which electrodes are surgically implanted permanently in the brain to modulate brain networks and function. In cervical dystonia, DBS of the postero-ventral part of the internal globus pallidus (GPi-DBS) has been established as an effective treatment for severe cases. However, the outcome of GPi-DBS in cervical dystonia has been reported mostly in some smaller series with up to 3 years follow-up. Thus, there is a lack of documentation of outcome of GPi-DBS in CD beyond 3 years of treatment and in larger patient materials. In this study the investigators will perform a long-term follow-up study of patients who were operated with a DBS-device targeting the GPi bilaterally, and who have been treated with chronic GPi-DBS for a minimum of 3 years. The investigators will measure the severity of symptom burden and quality of life with validated rating scales.

The investigators will compare this DBS-treated cohort with an age- and gender matched group of CD patients who are receiving the standard treatment with botulinum neurotoxin (BoNT) injections and have been treated for at least 3 years as well. The investigators hypothesize that the DBS-treated group will have a significantly lower burden of symptoms at long-term follow-up than the BoNT treated group.

DETAILED DESCRIPTION:
Cervical dystonia (CD) is the most common isolated dystonia in adults, with a prevalence of 9-13/100000. CD has a mean age at onset of 40 years, and is almost twice as common in women than in men. Cervical dystonia symptoms can in most patients be managed well by botulinum toxin (BoNT) injections, and supporting treatment measures. However, one-fifth to one-third of patients do not obtain sufficient relief from long-term BoNT therapy, resulting in reduced quality of life. Deep brain stimulation in the postero-ventral part of the internal globus pallidus (GPi-DBS) has been established as an effective treatment of cervical dystonia, including as a part of primary generalized dystonia, segmental or focal dystonia.

Long-term outcome of pallidal DBS in cervical dystonia has only been published in some smaller series. In a prospective, single-center study with blinded outcome assessments of eight CD patients, an average improvement of 70% in the Severity score of the TWSTRS , and 91% and 92% improvement, respectively, in the Disability and Pain scores, was found at median 30 months follow-up (Skogseid IM et al, 2012). The two largest unblinded series showed average improvements of TWSTRS Severity score of 55 % and 58 %, at mean follow-up 32 months (n=10), and 2 years (n=6), respectively (Hung SW et al, 2007, Cacciola F et al, 2010).

Although these studies are promising, there is a lack of documentation of outcome of GPi-DBS in CD beyond 3 years of treatment and in larger patient materials. Also, studies are lacking that compare the severity of remaining CD symptoms and disease-specific quality of life between a long-term treated DBS-cohort and a cohort receiving long-term BoNT treatment.

The investigators will therefore perform a cross-sectional, observational study of patients who were operated at Oslo University Hospital with a Medtronic DBS-device targeting the GPi bilaterally from 2004 to 2017, and who have been treated with chronic GPi-DBS for a minimum of 3 years and up to 13 years. The main objective is to assess remaining CD severity and CD-related Quality of Life (QoL) in this DBS-treated group and compare this with an age- and gender matched group of CD-patients treated with BoNT-injections for a minimum of 3 years (BoNT-group).

The main outcome measures are the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS), with its three subscores: Severity, Disability and Pain, and the Cervical Dystonia Impact Profile-58 (CDIP-58), which is a self-rated questionnaire for disease-specific quality of life. The primary endpoint of the study is the difference in TWSTRS total score between the two treatment groups at the time of long-term follow-up. The BoNT-group will be assessed with TWSTRS both before and 4-6 weeks after the last injection, but the score 4-6 weeks after injection will be used for comparison with the DBS-group. In the DBS-group the TWSTRS total and subscores obtained at long-term evaluation will also be compared to the scores which were obtained prior to the operation as part of the routine work-up. Secondary endpoints are TWSTRS Severity, Disability and Pain score, and CDIP-58 Total scores. Exploratory variables are the eight Symptom/Domain scores of the CDIP-58 and Visual Analog Scale for Global Burden of Disease (VAS-GBD), at long-term follow-up. Other outcome variables are complications and severe adverse events of the two treatment types, and the Anxiety and Depression scores of the Hospital Anxiety and Depression Scale (HADS).

The investigators hypothesize that the DBS-treated group will have a significantly lower mean TWSTRS total score at long-term follow-up than the BoNT treated group.

ELIGIBILITY:
Inclusion Criteria:

* DBS-group: Patients with isolated cervical dystonia (focal or part of segmental dystonia) who have been operated at Oslo University between June 2004 and June 2017 and treated with bilateral GPi-DBS for a minimum of 3 years, and who give their informed consent to participate in this follow-up study.
* BoNT-group: Patients who are receiving regular BoNT-injections at Oslo University Hospital for isolated cervical dystonia (focal or part of segmental dystonia), who are gender-and age-matched to the operated patients, and who give their informed consent to participate in this follow-up study.

Exclusion Criteria:

* Dementia/inability to respond to the CDIP-58.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have cervical dystonia, focal or segmental, and who have been receiving either GPi-DBS, or Botulinum toxin injections, for a minimum of 3 years, and who still receives such treatment. All patients to be included give their written informed consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Total score of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS). | In the DBS-group: After 3-17 years of continuous GPi-DBS. In the BoNT-group: After minimum 3 years of regular BoNT injections (minimum 12 injection cycles), and 4-6 weeks after the last injection.
  The TWSTRS is a validated clinical scale that assesses cervical dystonia symptom severity, disability and pain (Consky et al, 1990; Consky and Lang 1994; Comella et al, 1992; Dubinsky et al, 1991). In the first part the physical signs of cervical dystonia are scored by the investigator (Severity subscale), the second part rates disability/limitation of activities (Disability subscale), and the third part rates the intensity and duration of pain related to the CD, and its impact on the patient´s ability to participate in normal activities (Pain subscale).
  The TWSTRS Total score is the sum of the TWSTRS Severity score (0-35), the TWSTRS Disability score (0-30) and the TWSTRS Pain score (0-20), with a maximum total score of 85. Higher scores indicate more severe symptoms/disability/pain.

SECONDARY OUTCOMES:
Severity, Disability and Pain subscores of the TWSTRS | In the DBS-group: After 3-17 years of continuous GPi-DBS. In the BoNT-group: After minimum 3 years of regular BoNT injections (minimum 12 injection cycles),and 4-6 weeks after the last injection.
  The TWSTRS is a validated clinical scale that assesses cervical dystonia symptom severity, disability and pain (Consky et al, 1990; Consky and Lang 1994; Comella et al, 1992; Dubinsky et al, 1991). In the first part the physical signs of cervical dystonia are scored by the investigator (Severity subscale), the second part rates disability/limitation of activities (Disability subscale), and the third part rates the intensity and duration of pain related to the CD, and its impact on the patient´s ability to participate in normal activities (Pain subscale).
  The TWSTRS Total score is the sum of the TWSTRS Severity score (0-35), the TWSTRS Disability score (0-30) and the TWSTRS Pain score (0-20), with a maximum total score of 85. Higher scores indicate more severe symptoms/disability/pain.
Total score of the Cervical Dystonia Impact Profile 58 (CDIP-58) | In the DBS-group: After 3-17 years of continuous GPi-DBS. In the BoNT-group: After minimum 3 years of regular BoNT injections (minimum 12 injection cycles), and 4-6 weeks after the last injection.
  CDIP-58 is a patient-rated questionnaire that assesses disease-specific health-related quality of life. It includes 58 items grouped into eight dimensions. Summary scores of the eight dimensions are generated by summing items and are then transformed to a 0-100 scale. High scores indicate worse health.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Marie Skogseid, MDPhD, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- See also: Oslo University Hospital, homepage for Movement Disorders Research Group/Inger Marie Skogseid — https://www.ous-research.no/skogseid